CLINICAL TRIAL: NCT01728233
Title: Phase II Study of the Pan-HER Inhibitor Dacomitinib (PF-00299804) for Patients With Locally Advanced or Metastatic Squamous Cell Carcinoma of the Penis.
Brief Title: Dacomitinib (PF-00299804) in Advanced/Metastatic Squamous Cell Carcinoma of the Penis
Acronym: HER-Uro01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Andrea Necchi, MD, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT110/12
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Penile Neoplasms; Carcinoma, Squamous Cell
Keywords: Molecular Targeted Therapy; Neoadjuvant therapy; Dacomitinib
MeSH Terms: conditions — Penile Neoplasms; Carcinoma, Squamous Cell | interventions — dacomitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dacomitinib (PF-00299804) (Experimental): PF-299804 will be administered orally at a dose of 45 mg/day continuously until surgery, evidence of disease progression or onset of unacceptable toxicity.
  Interventions: Drug: Dacomitinib

INTERVENTIONS:
Drug: Dacomitinib — PF-299804 will be administered orally at a dose of 45 mg/day continuously until surgery, evidence of disease progression or onset of unacceptable toxicity.
  Other Names: PF-00299804

SUMMARY:
Penile squamous cell carcinoma (SCC) is a very rare disease and prognosis depends primarily on regional lymph-node involvement. Despite the fact that cure can be obtained in patients with low metastatic load (pN1) by monotherapy, combination therapy is required for more advanced cases. Medical treatment options only for advanced or metastatic penile SCC are not very effective so far and the few chances for cure are solely dependent on multimodality treatment, either with surgery or radiation. Based on the observation that the epidermal growth factor receptor (EGFR) is almost invariably expressed in penile SCC and assuming similarities to the SCC of head and neck district, anti-EGFR targeted monotherapy has been investigated with promising early results at Istituto Tumori Milan and University of Texas MD Andreson Cancer Center. These premises lend support to the use of the pan-HER inhibitor dacomitinib for advanced or metastatic penile SCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent
* Eastern Cooperative Oncology Group performance status of at least 1
* Cytologically or histologically proven diagnosis of SCC of the penis
* Uni- or bidimensionally measurable disease as defined by RECIST v1.1 criteria
* Clinical stage N2-3 and/or M1 (TNM 2002)
* Locoregional relapse after prior major surgery/ies (either single or multiple)
* No prior systemic therapy except for the administration of vincristine-bleomycin-methotrexate (VBM) chemotherapy for superficial disease if administered at least 6 months prior to study enrollment
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Central nervous system (CNS) metastases or leptomeningeal carcinomatosis
* History of active serious cardiovascular, cerebrovascular, pulmonary co-morbidities
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma or any cancer curatively treated > 5 years prior to study entry.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06-15 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the assessment of response-rate (RR) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. | 2-months
  RR (%) = complete response (CR) + partial response (PR), where CR is the disappearance of all target lesions (any pathological lymph-nodes must have reduction in short axis to < 10 mm) and PR indicates at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
To assess the safety and tolerability of the study drug. Incidence, nature and severity of treatment-related adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) v4.0. | 2-months
Pathologic complete response (pCR) rate for patients undergoing surgery in the treatment time course. | 2-months or longer.
Progression-free survival. | 2-months.
Overall Survival | 6-months
Variations of the Quality of Life score as assessed with the Edmonton Symptom Assessment Scale (ESAS), validated in Italian language. | 2-months.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Necchi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano; Roberto Salvioni, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy